CLINICAL TRIAL: NCT05039177
Title: A Phase 1b/2 Study of Agents Targeting the Mitogen-Activated Protein Kinase Pathway in Patients With Advanced Gastrointestinal Malignancies (HERKULES-3)
Brief Title: A Study of ERAS-007 in Patients With Advanced Gastrointestinal Malignancies
Acronym: HERKULES-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-007-03
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: BRAF; V600E; KRAS; NRAS; mutation; Braftovi; encorafenib; Erbitux; cetuximab; Ibrance; palbociclib; ERK; MAPK; CDK4/6; CRC; colorectal cancer; EGFR; GI neoplasm; gastrointestinal neoplasm; PDAC; Pancreas Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms | interventions — encorafenib; Cetuximab; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Parts A1a, A2a, or A3a): ERAS-007 in combination with encorafenib and cetuximab (Experimental): ERAS-007 will be orally administered in combination with encorafenib and cetuximab to study participants with BRAFm CRC in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: Encorafenib; Drug: Cetuximab
- Dose Escalation (Parts B1a, B2a, B3a or B4a): ERAS-007 in combination with palbociclib (Experimental): ERAS-007 will be orally administered in combination with palbociclib to study participants with KRASm or NRASm CRC and KRASm PDAC in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: Palbociclib
- Dose Expan (Parts A1b, A1c, A2b, A2c, A3b, or A3c): ERAS-007 in combo with encorafenib & cetuximab (Experimental): ERAS-007 will be orally administered at the recommended dose (as determined from Parts A1a, A2a or A3a) in combination with encorafenib and cetuximab to study participants with BRAFm CRC.
  Interventions: Drug: ERAS-007; Drug: Encorafenib; Drug: Cetuximab
- Dose Expansion (Parts B1b, B2b, B3b, and B4b): ERAS-007 in combination with palbociclib (Experimental): ERAS-007 will be orally administered at the recommended dose (as determined from Parts B1a, B2a, B3a or B4a) in combination with palbociclib to study participants with KRASm or NRASm CRC.
  Interventions: Drug: ERAS-007; Drug: Palbociclib

INTERVENTIONS:
Drug: ERAS-007 — Administered orally
Drug: Encorafenib — Administered orally
  Other Names: Braftovi
  Arms: Dose Escalation (Parts A1a, A2a, or A3a): ERAS-007 in combination with encorafenib and cetuximab; Dose Expan (Parts A1b, A1c, A2b, A2c, A3b, or A3c): ERAS-007 in combo with encorafenib & cetuximab
Drug: Cetuximab — Administered via intravenous infusion
  Other Names: Erbitux
  Arms: Dose Escalation (Parts A1a, A2a, or A3a): ERAS-007 in combination with encorafenib and cetuximab; Dose Expan (Parts A1b, A1c, A2b, A2c, A3b, or A3c): ERAS-007 in combo with encorafenib & cetuximab
Drug: Palbociclib — Administered orally
  Other Names: Ibrance
  Arms: Dose Escalation (Parts B1a, B2a, B3a or B4a): ERAS-007 in combination with palbociclib; Dose Expansion (Parts B1b, B2b, B3b, and B4b): ERAS-007 in combination with palbociclib

SUMMARY:
* To evaluate the safety and tolerability of escalating doses of ERAS-007 in combination with other cancer therapies in study participants with advanced GI malignancies.
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-007 administered in combination with other cancer therapies.
* To evaluate the antitumor activity of ERAS-007 in combination with other cancer therapies.
* To evaluate the PK profiles of ERAS-007 and other cancer therapies when administered in combination.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, multicenter clinical study evaluating ERAS-007 in combination with other cancer therapies in study participants with GI malignancies. This study will serve as a platform study, allowing for evaluation of safety/tolerability and efficacy of ERAS-007 in combination with other cancer therapies. The study will initially commence with dose escalation of ERAS-007 administered in combination with encorafenib and cetuximab in study participants with metastatic colorectal cancer (CRC) harboring B-Raf proto-oncogene, serine/threonine kinase (BRAF) V600E mutation; and dose escalation of ERAS-007 administered in combination with palbociclib in study participants with metastatic CRC harboring Kirsten rat sarcoma (KRAS) or neuroblastoma rat sarcoma (NRAS) mutations and metastatic pancreatic adenocarcinoma with (PDAC) KRAS mutation. Dose expansion will follow and will test ERAS-007 administered at the RD identified from each dose escalation arm in study participants with metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willing and able to give written informed consent.
* Have histologically or cytologically confirmed metastatic CRC harboring applicable mutation(s) (e.g., BRAF V600E; KRAS or NRAS mutations) or metastatic PDAC harboring KRAS mutation based on an analytically validated assay performed on tumor tissue in a certified testing laboratory.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Adequate bone marrow and organ function.
* Have ECOG performance status of 0 or 1.
* Willing to comply with all protocol-required visits, assessments, and procedures.
* Able to swallow oral medication.

Exclusion Criteria:

* Prior therapy with a RAS, MEK, or ERK inhibitor. Depending on which treatment arm the patient is assigned, other therapies could also be prohibitive.
* Anti-cancer therapy ≤ 21 days or 4 half-lives prior to first dose of study drug, whichever is shorter.
* Palliative radiation ≤ 7 days prior to first dose of study drug.
* Symptomatic brain metastasis or leptomeningeal disease.
* Gastrointestinal conditions that may affect absorption of oral medications
* Active infection requiring systemic therapy, or a known history of HIV infection, hepatitis B virus, or hepatitis C virus.
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months prior to first study drug dose.
* Active, clinically significant interstitial lung disease or pneumonitis.
* Impaired cardiovascular function or clinically significant cardiovascular disease.
* History of thromboembolic or cerebrovascular events ≤ 6 months prior to first dose.
* Major surgery within 28 days of enrollment, or anticipation of major surgery during study treatment.
* Known intolerance or contraindication to encorafenib, cetuximab, or palbociclib.
* Pregnant or breastfeeding women.
* Any evidence of severe or uncontrolled systemic disease or evidence of any other significant clinical disorder or laboratory finding that renders the patient inappropriate to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Maximum Tolerated Dose (MTD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Recommended Dose (RD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma or serum concentration of ERAS-007 and other cancer therapies
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma or serum concentration of ERAS-007 and other cancer therapies
Area under the curve | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve of ERAS-007 and other cancer therapies
Half-life | Study Day 1 up to Day 29
  Half-life of ERAS-007 and other cancer therapies
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Antal, Study Director — Clinical Development
Locations (14):
- United States (14):
  - University of Alabama at Birmingham (O'Neal Comprehensive Cancer Center), Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California Irvine College of Medicine, Orange, California
  - UCSF Mount Zion Medical Ctr, San Francisco, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University (Siteman Cancer Center), St Louis, Missouri
  - Duke Cancer Institute, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No